CLINICAL TRIAL: NCT06887608
Title: The Effect of Partner-Assisted Rebozo Application in the Intrapartum Period on Birth Fear, Pain and Satisfaction
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, dilan cömert, Phd Candidate, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 27.01.2025-1187899
Record Dates: First submitted 2025-03-16; First posted 2025-03-20 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-06

CONDITIONS: Rebozo at Birth
Keywords: birth, rebozo, fear of birth, birth pain, satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: It was designed as a randomized controlled experimental study.
Who Masked: Participant
Masking Description: In order to increase the reliability of the research and to distribute the groups homogeneously, groups will be assigned from the website www.randomizer.org. Pregnant women belonging to all three groups will be assigned to the groups through this website.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- husband supported rebozo group (Experimental): In the partner-assisted rebozo group, information will be provided to the partner and the pregnant woman with the education booklet created during the latent phase and training will be provided. When the pregnant woman reaches 4-5 cm, 6-7 cm and 8-9 cm vaginal dilation, the data collection forms and scale forms determined for the pregnant woman in the partner-assisted rebozo group will be filled in before the rebozo application. Rebozo application will be applied to the pregnant woman for three contractions. A re-evaluation will be made after the rebozo application. The determined scales will be applied at the 4th hour in the postpartum period.
  Interventions: Other: Husband assisted rebozo application
- midwife assisted rebozo group (Experimental): In the midwife-assisted rebozo group, information will be provided to the pregnant woman with the education booklet created during the latent phase and training will be provided. When the pregnant woman reaches 4-5 cm, 6-7 cm and 8-9 cm vaginal dilation, the data collection forms and scale forms determined for the pregnant woman in the midwife-assisted rebozo group will be filled in before the rebozo application. Rebozo application will be applied to the pregnant woman for three contractions. A re-evaluation will be made after the rebozo application. The determined scales will be applied at the 4th hour in the postpartum period.
  Interventions: Other: Midwife assisted rebozo application
- control group (No Intervention): In the control group, when the pregnant woman reaches 4-5 cm, 6-7 cm and 8-9 cm vaginal opening, the same measurements will be made and the woman will continue to receive routine care, and then the measurements will be repeated. In the 4th hour after birth, the determined scales will be applied.

INTERVENTIONS:
Other: Husband assisted rebozo application — At 4-5 cm, 6-7 cm and 8-9 cm, the pregnant woman will be given a rebozo by her husband.
  Arms: husband supported rebozo group
Other: Midwife assisted rebozo application — The midwife will apply rebozo to the pregnant woman at 4-5 cm, 6-7 cm and 8-9 cm.
  Arms: midwife assisted rebozo group

SUMMARY:
The World Health Organization (WHO) recommends the use of non-pharmacological methods for the relief of labor pain. The use of non-pharmacological methods in pain management helps women see their labor as a natural event and contributes to the reduction of cesarean section rates by increasing satisfaction with normal birth . The rebozo technique, a traditional method, originates from Latin America and is a non-invasive, non-drug practical application. The rebozo technique reduces or eliminates pain by creating rhythmic movements in the pelvic area. No study has been found evaluating the results of partner-assisted rebozo application in the intrapartum period. For this reason, it is important to conduct evidence-based studies examining the effects of the use of rebozo technique in labor. This randomized controlled study will contribute to the literature. For this purpose, this study was planned to examine the effects of partner-assisted rebozo application in the intrapartum period on fear of labor, pain, and labor satisfaction.

DETAILED DESCRIPTION:
Childbirth is a challenging and life-changing experience for women that has emotional and physical effects. Every woman wants to remember her childbirth as a positive process, but the pain and suffering that accompanies this process can affect the perception of the pregnant woman. A long labor can increase complications for the baby and the mother. Despite all this, adapting to labor pain increases women's satisfaction with the labor process. For this, it is necessary to adopt methods that can reduce the duration and intensity of labor pain to a safe range and thus facilitate adaptation to pain. The American College of Obstetricians and Gynecologists (ACOG) recommends appropriate interventions to relieve labor pain. The World Health Organization (WHO) recommends the use of non-pharmacological methods for the relief of labor pain. The use of non-pharmacological methods in pain management helps women see their birth as a natural event and increases satisfaction with normal birth, thus contributing to the reduction of cesarean section rates. The rebozo technique, a traditional method, originates from Latin America and is a non-invasive, non-drug practical application. The rebozo technique reduces or eliminates pain levels by creating rhythmic movements in the pelvic area. Rebozo can be used before, during and after birth. When applied during labor, it corrects fetal malpositions, allows the fetus to easily make cardinal movements, and accelerates the progression of labor. There are limited studies on the rebozo application in the literature. In studies, women stated that they relaxed during contractions and their attention shifted away from the pain. In Febby's (2019) study, it was stated that the mother felt more comfortable with the rebozo technique, that it caused a hug-like feeling in the mother, causing the release of oxytocin, which could make the birth process faster and less painful, and that it could increase the sense of comfort among mothers. In a qualitative study, it was reported that pregnant women felt physically good with the application of the rebozo technique, that it was effective in reducing pain, and that especially when applied by midwives, it created great satisfaction in the mother. The application of the technique by midwives during labor will ensure that the pregnant woman actively participates in the labor, establishes a relationship of trust between the midwife and the pregnant woman, helps the pregnant woman cope with the pain of labor, and increases satisfaction with the labor. In the literature, it has been determined that rebozo application in the active phase reduces anxiety level and pain score and increases satisfaction. In a study, it was stated that the rebozo technique increases the rate of fetal descent and cervical dilatation. In another study, it was determined that the length of the second stage of labor with the rebozo technique was 27.07 minutes shorter than the control group. There are limited clinical studies conducted in our country with the rebozo technique. There is no study evaluating the results of partner-assisted rebozo application in the intrapartum period. For this reason, it is important to conduct evidence-based studies examining the effects of the use of rebozo technique in labor. This randomized controlled study will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being literate,
* Knowing Turkish,
* Being over 18 years of age,
* Being primiparous,
* Having a single fetus and cephalic presentation,
* Being at term (37-42 weeks),
* Not having risk factors during pregnancy (Preeclampsia, premature rupture of membranes, oligohydramnios and polyhydramnios, gestational diabetes, placental anomalies, intrauterine growth retardation, intrauterine dead fetus, fetal distress, macrosomic babies, etc.),
* Being in the active phase of the first stage of labor,
* Those who agree to participate in the research,
* The spouse also agrees to participate in the research.

Exclusion Criteria:

* Being multiparous,
* Having multiple pregnancies,
* Women with any chronic disease,
* Women with a diagnosed psychiatric disease,
* Pregnant women with spine and bone structure problems.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who are coming to birth and are 4-5 cm dilated in their first pregnancy
Enrollment: 120 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 8 hours
  Visual analog scale (VAS): The pain levels of the participants will be evaluated with the Visual analog scale (VAS). It was developed by Bond and Pilowski in 1966 in order to describe the severity of pain in individuals numerically. This measurement tool is a 10 cm long ruler. While the expression "no pain" is written on the left end, the expression "unbearable pain" is written on the right end. Since it has linear properties, the difference between each increase is equal. It is the most commonly used single-dimensional scale type because it does not guide individuals with numbers due to its usage feature, the evaluation is easy and fast, and it gives results in a short time. A VAS value approaching 10 indicates that the pain is very severe, while a value approaching 0 is evaluated as the pain has decreased.
Birth Satisfaction Scale: | 8 hours
  Birth Satisfaction Scale: Participants' satisfaction levels will be assessed with the Birth Satisfaction Scale. The scale, which was developed to assess women's perceptions of birth, was developed by Martin and Fleming in 2009. Its Turkish validity and reliability were made by Çoşar Çetin and colleagues in 2015. The scale is Likert-type and is scored from 5 (Strongly agree) to 1 (Strongly disagree). Items 4, 8, 12, 15, 16, 17, 19, 20, 21, 23, 25, and 29 are scored reversely. The scale has 30 items and the possible score varies between 30-150. There is no cut-off point for the scale. As the score increases, satisfaction with birth increases. The scale has 3 sub-dimensions: Quality of care (home assessment, birth environment, adequate support and communication with healthcare personnel), personal characteristics of women (ability to cope with birth, sense of control, preparation for birth, communication with the baby), and stress experienced during the birth process (experiencing distre
Fear of Childbirth Scale: | 8 hours
  Fear of Childbirth Scale: Participants' fear levels will be assessed with the Fear of Childbirth Scale. The scale measures fear during childbirth. The scale, developed by Wijma et al. (2002), was validated in Turkish by Serçekuş et al. in 2017 for validity and reliability. The scale measuring fear during childbirth consists of 10 items. The scale takes 30-90 seconds to administer. Each item in the scale is asked to be scored from 1 (completely disagree) to 10 (completely agree). The possible scores from the scale are between 10-100. A high score indicates high fear. It is an extremely practical scale in terms of application. 5 items (1,3,5,7,10) in the scale are positive and 5 items (2,4,6,8,9) are negative. The 5 items with positive meanings on the scale are reverse scored. The scale can be applied to all multiparous and primiparous women who are admitted to the delivery room and have cervical dilatation of 3 cm or more. The Cronbach alpha reliability coefficient of the scale is 0.88

CONTACTS AND LOCATIONS:
Overall Officials: DİLAN C Phd Candidate, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul Training and Research Hospital, Zeytinburnu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No